CLINICAL TRIAL: NCT05144698
Title: Phase I/II Trial of Autologous Rapamycin-Resistant Th1/Tc1 (RAPA-201) Cell Therapy of PD-(L)1 Resistant Solid Tumors
Brief Title: RAPA-201 Therapy of Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rapa Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPA-201-STP-01
Record Dates: First submitted 2021-11-05; First posted 2021-12-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor; Small Cell and Non-small Cell Lung Cancer; Head and Neck Cancer; Squamous Cell Carcinoma of Oral Cavity; Squamous Cell Carcinoma of Larynx; Squamous Cell Carcinoma of Nasopharynx; Squamous Cell Carcinoma of Other Specified Sites of Skin; Malignant Melanoma; Esophageal Squamous Cell Carcinoma
Keywords: Refractory to Checkpoint Therapy; PD-1; PD-L1; Adoptive T cell therapy; Regenerative Medicine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Non-randomized, open label, multi-site, phase I/II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of RAPA-201 cells (Experimental): RAPA-201 cells will be administered at a target flat dose of 400 x 10^6 cells per infusion. After RAPA-201 therapy, anti-PD1 maintenance therapy (pembrolizumab, 200 mg administered intravenously every 3 weeks for up to 12 months)
  Interventions: Biological: RAPA-201 Rapamycin Resistant T Cells; Drug: Chemotherapy Prior to RAPA-201 Therapy; Drug: Pembrolizumab (PD-1 Blocking Antibody)

INTERVENTIONS:
Biological: RAPA-201 Rapamycin Resistant T Cells — Autologous Rapamycin-Resistant Th1/Tc1 Cells
  Other Names: RAPA-201 cells
Drug: Chemotherapy Prior to RAPA-201 Therapy — Outpatient Carboplatin + Paclitaxel Regimen (CP Regimen)
Drug: Pembrolizumab (PD-1 Blocking Antibody) — Drug Therapy After RAPA-201 Therapy

SUMMARY:
The therapy of solid tumors has been revolutionized by immune therapy, in particular, approaches that activate immune T cells in a polyclonal manner through blockade of checkpoint pathways such as PD-1 by administration of monoclonal antibodies. In this study, the investigators will evaluate the adoptive transfer of RAPA-201 cells, which are checkpoint-deficient polyclonal T cells that represent an analogous yet distinct immune therapy treatment platform for solid tumors. The administration of polyclonal, metabolically-fit RAPA-201 cells is a novel adoptive T cell therapy approach that is suitable for regenerative medicine efforts.

RAPA-201 is a novel immunotherapy product consisting of reprogrammed autologous CD4+ and CD8+ T cells of Th1/Tc1 cytokine phenotype. RAPA-201, which have acquired resistance to the mTOR inhibitor temsirolimus, are manufactured ex vivo from peripheral blood mononuclear cells collected from solid tumor patients using a steady-state apheresis. The novel RAPA-201 manufacturing platform, which incorporates both an mTOR inhibitor (temsirolimus) and an anti-cancer Th1/Tc1 polarizing agent (IFN-alpha) generates polyclonal T cells with five key characteristics:

1. Th1/Tc1: polarization to anti-cancer Th1 and Tc1 subsets, with commensurate down-regulation of immune suppressive Th2 and regulatory T (TREG) subsets;
2. T Central Memory: expression of a T central memory (TCM) phenotype, which promotes T cell engraftment and persistence for prolonged anti-tumor effects;
3. Rapamycin-Resistance: acquisition of rapamycin-resistance, which translates into a multi-faceted anti-apoptotic phenotype that improves T cell fitness in the stringent conditions of the tumor microenvironment;
4. T Cell Quiescence: reduced T cell activation, as evidence by reduced expression of the IL-2 receptor CD25, which reduces T cell-mediated cytokine toxicities such as cytokine-release syndrome (CRS) that limit other forms of T cell therapy; and
5. Reduced Checkpoints: multiple checkpoint inhibitory receptors are markedly reduced on RAPA-201 cells (including but not limited to PD-1, CTLA4, TIM-3, LAG3, and LAIR1), which increases T cell immunity in the checkpoint-replete, immune suppressive tumor microenvironment.

This is a non-randomized, open label, multi-site, phase I/II trial of outpatient RAPA-201 immune T cell therapy in patients with advanced metastatic, recurrent, and unresectable solid tumors that have recurred or relapsed after prior immune therapy. Patients must have tumor relapse after at least one prior line of therapy and must have refractory status to the most recent regimen, which must include an anti-PD-(L)1 monoclonal antibody. Furthermore, accrual focuses upon solid tumor disease types potentially amenable to standard-of-care salvage chemotherapy consisting of the carboplatin + paclitaxel (CP) regimen that will be utilized for host conditioning prior to RAPA-201 therapy. Importantly, carboplatin and paclitaxel are "immunogenic" chemotherapy agents whereby the resultant cancer cell death mechanism is favorable for generation of anti-tumor immune T cell responses. Thus, the CP regimen that this protocol incorporates is intended to directly control tumor progression and indirectly promote anti-tumor T cell immunity.

Protocol therapy consists of six cycles of standard-of-care chemotherapy (carboplatin + paclitaxel (CP) regimen) administered in the outpatient setting every 28 days (chemotherapy administered on cycles day 1, 8, and 15). RAPA-201 cells will be administered at a target flat dose of 400 X 10^6 cells per infusion on day 3 of cycles 2 through 6.

In the original protocol design, a sample size of up to 22 patients was selected to determine whether RAPA-201 therapy, when used in combination with the CP regimen, represents an active regimen in solid tumors that are resistant to anti-PD(L)-1 checkpoint inhibitor therapy, as defined by a response rate (≥ PR) consistent with a rate of 35%. The first stage of protocol accrual consisted of n=10 patients; to advance to the second protocol accrual stage (accrual of an additional n=12 patients), RAPA-201 therapy must result in a tumor response (≥ PR) in at least 2 out of the 10 initial patients. As described below in the detailed description, this original protocol implementation demonstrated that RAPA-201 represented an active treatment regimen for solid tumor patients, and as such, the protocol was expanded to evaluate the combination of RAPA-201 therapy followed by anti-PD1 maintenance therapy.

DETAILED DESCRIPTION:
The therapy of solid tumors has been revolutionized by immune therapy, in particular, approaches that activate immune T cells in a polyclonal manner through blockade of checkpoint pathways such as PD-1 by administration of monoclonal antibodies. In this study, the investigators will evaluate the adoptive transfer of a reprogrammed T cell population termed RAPA-201 cells, which are checkpoint-deficient polyclonal T cells that represent an analogous yet distinct treatment platform for solid tumor immune therapy.

RAPA-201 is a novel T cell immunotherapy product that is comprised of autologous CD4+ and CD8+ T cells of Th1/Tc1 cytokine phenotype. The RAPA-201 cells, which have acquired resistance to the mTOR inhibitor temsirolimus, are manufactured ex vivo from peripheral blood mononuclear cells collected from solid tumor patients using a steady-state apheresis. RAPA-201 cells are also being evaluated for the therapy of relapsed, refractory multiple myeloma and was granted Fast Track Status by the FDA for this indication. The novel method of RAPA-201 manufacturing, which incorporates both an mTOR inhibitor (temsirolimus) and an anti-cancer Th1/Tc1 polarizing agent (IFN-alpha) generates a polyclonal T cell population with the following five key characteristics:

1. Th1/Tc1: polarization to the anti-cancer Th1 and Tc1 subsets, with commensurate down-regulation of immune suppressive Th2 and regulatory T (TREG) subsets;
2. T Central Memory: expression of a T central memory (TCM) phenotype, which promotes T cell engraftment and persistence necessary for prolonged anti-tumor effects;
3. Rapamycin-Resistance: acquisition of rapamycin-resistance, which translates into a multi-faceted anti-apoptotic phenotype that improves T cell fitness in the stringent conditions of the tumor microenvironment;
4. T Cell Quiescence: reduced T cell activation, as evidence by reduced expression of the IL-2 receptor CD25, which reduces the chance of T cell-mediated cytokine toxicities such as cytokine-release syndrome (CRS) that limit other forms of T cell therapy; and
5. Reduced Checkpoints: multiple checkpoint inhibitory receptors are markedly reduced on RAPA-201 cells (including but not limited to PD-1, CTLA4, TIM-3, LAG3, and LAIR1), which increases T cell immunity in the checkpoint-replete, immune suppressive tumor microenvironment.

This is a multi-site phase I/II study evaluating RAPA-201 cells in up to 22 patients with relapsed solid tumors who have disease progression after anti-PD1 pathway monoclonal antibody therapy. In the initial protocol implementation, which studied n=22 evaluable participants, patients with malignant melanoma, small cell lung cancer, non-small cell lung cancer, gastric cancer, and squamous cell head and neck cancer were accrued. RAPA-201 therapy caused iRECIST-defined partial responses in 10 of 22 patients, with responses in melanoma (6/10 PR, 60% response rate), small cell lung cancer (2/3 PR, 66% response rate), and head and neck cancer (2/3 responses, 66% response rate). On the basis of this significant response rate in metastatic, treatment-resistant malignant melanoma, RAPA-201 treatment for this disease indication was granted the Regenerative Medicine Advanced Therapeutics (RMAT) designation by the US FDA. Some patients with non-small cell lung cancer had a delay in time to progression relative to their previous treatment regimen. RAPA-201 therapy was also safely administered exclusively in the outpatient setting; specifically, there were no adverse events of any grade attributable to RAPA-201, including no cytokine release syndrome (CRS). Given these early signals of safety and efficacy, the protocol was amended to accrue n=15 additional participants. Given the phase 1 response data, the additional n=15 study participants will consist of patients with refractory melanoma, small cell lung cancer, squamous cell head and neck cancer, and non-small cell lung cancer. In addition, this expanded cohort of n=15 study participants will receive anti-PD1 monoclonal antibody maintenance therapy after RAPA-201 cell therapy (patients in the initial n=22 study cohort did not receive anti-PD1 maintenance). The study evaluates adoptive T cell therapy using autologous rapamycin-resistant Th1/Tc1 cells (RAPA-201) in the context of a standard-of-care chemotherapy regimen comprised of carboplatin plus paclitaxel (CP Regimen), which is considered "immunogenic" chemotherapy whereby the resultant cancer cell death mechanism is favorable for the generation of anti-tumor immune T cell responses. Therefore, the CP regimen that this protocol incorporates is intended to both directly control tumor progression and indirectly promote anti-tumor T cell immunity.

To be eligible for the protocol, a subject will be required to have a circulating absolute lymphocyte count (ALC) of ≥ 300 cells per microliter. This parameter will help ensure that a sufficient number of autologous RAPA-201 cells can be manufactured from a steady-state apheresis product. Once the apheresis product has been received at the manufacturing site, the subject can initiate the first cycle of the CP Regimen, which will be administered over a 28-day interval.

Within 10 days after positive determination of study eligibility (and subject enrollment), two key actions will occur: (1) T cells will be collected by steady-state apheresis and sent to the manufacturing site at Rapa Therapeutics; (2) and the patient will start Cycle 1 of the CP Regimen (with a window of up to 7 calendar days to begin).

The Carboplatin-Paclitaxel (CP) regimen will be given alone for Cycle 1 and in combination with RAPA-201 cells for Cycles 2-6. After the completion of the treatment portion of the study, the subject will enter the follow-up component that will last for 6 months.

Cycle 1 of the CP Regimen will be a 28-day cycle, which will allow for time to manufacture the RAPA-201 cell product. According to standard-of-care practice, the carboplatin and paclitaxel will be administered on days 1, 8, and 15 of each cycle. Each cycle, beginning with Cycle 1, may be delayed or extended for up to four weeks, if needed for various reasons, including: logistical considerations, resolution of adverse events, or if there is a delay in RAPA-201 manufacturing. Requests for using additional time between cycles, other than the visit windows specified in the Schedule of Events, should be approved by the Medical Monitor.

Cycles 2-6 will also be 28-day cycles but will include the infusion of RAPA-201 cells at a target flat dose of 400 X 10^6 cells per infusion (administered on day 3 of the CP regimen).

A sample size of n= 15 patients in the amended protocol design was selected to evaluate the safety and potential beneficial ant-tumor effect RAPA-201 therapy plus anti-PD1 maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
3. Advanced metastatic, recurrent, and unresectable solid tumor that has relapsed after ≥ one prior line of therapy.
4. Subject must have received prior therapy with disease-specific regimens that have been established to convey a clinical benefit. Alternatively, subject must have been offered such regimens and provided written documentation of refusal to receive such regimens.
5. Subject with solid tumors with genetic alterations and mutations (including but not limited to BRAF, BRCA, EGFR mutations, and ALK translocations) must have either received targeted therapy for such conditions or provided written documentation of refusal to receive such regimens.
6. Exposure to an anti-PD-(L)1 monoclonal antibody therapeutic in the most recent line of prior therapy.
7. Documented refractory status to the most recent regimen, which must include an anti-PD-(L)1 monoclonal antibody, as defined by lack of response after at least two cycles of therapy or relapse within 12-months of initiation of anti-PD-(L)1-containing therapy.
8. Solid tumor disease types that are eligible for enrollment consist of:

   1. head and neck cancer (squamous cell carcinoma of oral cavity, larynx, nasopharynx, and other sites);
   2. malignant melanoma;
   3. small cell carcinoma, thoracic and extra-thoracic; and,
   4. non-small cell lung cancer.
9. Presence of measurable disease to permit monitoring by RECISTv1.1 Criteria.
10. Must have a potential source of autologous T cells potentially sufficient to manufacture RAPA-201 cells, as defined by a circulating absolute lymphocyte count (ALC) of ≥ 300 cells/μL.
11. Patients must be ≥ two weeks from last solid tumor cancer chemotherapy, major surgery, radiation therapy and/or participation in investigational trials.
12. Patients must have recovered from clinical toxicities (resolution of CTCAE (v5) toxicity to a value of ≤ 2).
13. Ejection fraction (EF) by MUGA or 2-D echocardiogram within institution normal limits, with an EF level of ≥ 40%.
14. Calculated creatinine clearance of ≥ 60 mL/min/1.73 m^2.
15. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 x upper limit of normal.
16. ANC (Absolute neutrophil count) of ≥ 1500 cells/μL.
17. Platelet count ≥ 100,000 cells/μL.
18. Hemoglobin count ≥ 8 grams/μL.
19. Bilirubin ≤ 1.5 mg/dL (except if due to Gilbert's disease).
20. Corrected DLCO ≥ 50% (Pulmonary Function Test)
21. No history of abnormal bleeding tendency (as defined by any inherited coagulation defect, or history of internal bleeding).
22. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Other active malignancy (except non-melanoma skin cancer).
2. Life expectancy < 4 months.
3. Seropositivity for HIV, hepatitis B, or hepatitis C, unless such conditions are in stable condition using adequate treatment.
4. Uncontrolled hypertension.
5. History of cerebrovascular accident within 6 months of enrollment.
6. Myocardial infarction within 6 months prior to enrollment.
7. NYHA class III/IV congestive heart failure.
8. Uncontrolled angina/ischemic heart disease.
9. Cancer metastasis to the central nervous system, unless such metastasis has been adequately treated.
10. Pregnant or breastfeeding patients.
11. Patients of childbearing age, or males who have a partner of childbearing potential, who are unwilling to practice contraception.
12. Patients may be excluded at the discretion of the PI or if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the rate of Treatment Emergent Adverse Events of RAPA-201 using host conditioning of Carboplatin plus Paclitaxel | Completion of RAPA-201 Therapy plus combination anti-PD1 maintenance therapy; occurs on average at 18-months after treatment initiation
  To determine the safety of RAPA-201 cell therapy when used in combination with a carboplatin plus paclitaxel (CP) standard-of-care chemotherapy regimen and in combination with anti-PD1 maintenance therapy. Specifically, the treatment will be determined to be safe if the following parameters are met: (Metric #1) using the metric of "grade 4/grade 5 toxicity toxicity attributable to the RAPA-201 cell therapy": for positive determination of safety, this metric must occur in 1 or fewer patients out of the initial 10 patients.

SECONDARY OUTCOMES:
Overall Response Rate | One (1) year after the last dose of RAPA-201 cells.
  To determine the overall RECISTv1.1 criteria response rate (partial response or better) of autologous RAPA-201 cells and standard-of-care chemotherapy (carboplatin + paclitaxel) plus anti-PD1 maintenance therapy in patients with solid tumors resistant to PD-(L)1.
Progression Free Survival (PFS) and Overall Survival (OS) | One (1) year after the last dose of RAPA-201 cells.
  To characterize the effect of therapy on solid tumor disease control, as measured by progression free survival (PFS) and overall survival (OS).
Quality of Life (QOL) | One (1) year after the last dose of RAPA-201 cells.
  To evaluate effect of therapy on quality of life (QOL) using the Short Form-36 Survey.

OTHER OUTCOMES:
T Cell Immune Reconstitution | One (1) year after study start.
  To characterize the phenotype of immune T cell reconstitution, as defined by peripheral blood T cell count, which will be determined by flow cytometry using the CD3+ marker. CD3+ T cell count will be compared pre-treatment (at study entry) and at one-year after study start.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fowler, M.D., Study Director — Rapa Therapeutics LLC
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No